CLINICAL TRIAL: NCT07273669
Title: Advanced Robotic Beds for the Early Rehabilitation of Cardiac Surgery Patients
Acronym: CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Gennaro Galasso, Professor of cardiology, University of Salerno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PNRR-MCNT2-2023-12378283; PNRR-MCNT2-2023-12378283 (Other Grant/Funding Number: Ministero della Salute, Italian Health Ministry)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: AORTIC VALVE DISEASES; Mitral Valve Failure
Keywords: Robotic Beds; early rehabilitation; cardiac surgery; post cardiac surgery ICU
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of the robotic bed (Experimental): LOLE.K use
  Interventions: Device: use of the robotic bed
- Physicians standard of care (No Intervention)

INTERVENTIONS:
Device: use of the robotic bed — use of the robotic bed LOLE.K for the early rehabilitation
  Arms: Use of the robotic bed

SUMMARY:
The goal of this clinical trial is to evaluate whether LOLE.K, a new and specialized robotic bed, is effective in the rehabilitation of patients who have undergone surgery. The primary objectives of the trial are:

* Efficacy of LOLE.K: Does the LOLE.K robotic bed improve early rehabilitation in patients who undergone cardiac surgery?
* Impact on recovery: Does LOLE.K influence wound healing, muscle and neurological recovery, and psychological well-being?

To address these questions, the researchers will compare the use of LOLE.K with standard physical therapy to determine whether the robotic bed results in better outcomes in post-operative rehabilitation.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn whether LOLE.K, a new and specialized robotic bed, works for rehabilitation of patients following surgery.

The main research questions are:

1. Is LOLE.K effictive in enhancing early rehabilitation among patients who have undergone cardiac surgery?
2. Does LOLE.K influence wound healing, muscular and neurological recovery, and psychological well-being?

Researchers will compare LOLE.K bed to the usual therapy to see if LOLE.K woks better than standard post-operation rehabilitation.

1. Project Objectives Primary Objective: To assess the effectiveness of multirole robotic beds (LOLE.K) for early rehabilitation in cardiac surgery patients.
2. Target Population Patients: individuals aged 60-85 years undergoing aortic and mitral valve surgery.

   Study Sites: University of Salerno Hospital and IRCCS Ospedale Galeazzi-Sant'Ambrogio.
3. Experimental Design:

   * Control Group: Standard post-operative rehabilitation.
   * Experimental Group: Rehabilitation using LOLE.K robotic beds.
4. Key phases

   - Pilot Phase (Months 1-6): Define dataset structure, initiate patient enrollement and refine the operational algorithm.

   - Enrollment Phase (Months 6-12): Collect demographic, clinical, and physical health data from enrolled patients.

   - Follow-Up & Analysis Phase (Months 12-24): Perform in-depth statistical analysis and finalize outcome evalitaion.
5. Data Colection Data Types: Demographic, clinical, physical, echocardiographic, and wound-healing data.

   Devices: LOLE.K robotic beds and echography machines.
6. Outcomes & Measurements

   * Primary Outocomes: Lenght of hospital stay, ICU requirements, and rehabilitation time.
   * Secondary: Lung function, mental health scores, wound-healing scores, quality of life and cardiac output improvements.

   Standardized protocols for sedation and analgesia management will be applied, including the Richmond Agitation-Sedation Scale (RASS) for sedation and the Behavioral Pain Scale (BPS) or Critical Pain Observation Tool (CPOT) for pain. Also, delirium will be assessed using the Confusion Assessment Method for ICU (CAM-ICU). These parametres are critical: if patients are overly sedated or inadequately anesthetized, the results on mobilization could be confounded by these factors. Assessment of delirium is important because early mobilization could also have beneficial effects on cognitive status.
7. Statistical Analysis Plan

   * Descriptive Statistics: To provide an overview of baseline data.
   * Regression Models: To analyze the impact of key variables on clinical outcomes.
   * Machine Learning Models: To evaluate treatment efficiency based on patient data.
8. Expected Outcomes The use of LOLE.K is expected to result in faster recovery times, reduced ICU stays, improved physical and mental health, and enhanced wound healing compared with standard post-operative rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing aortic and mitral vale surgery
* patients aged between 60 and 85

Exclusion Criteria:

* Age < 18 years old
* inability to provide informed consent, either verbally or in writing, or unwillingness to participate in systematic follow-up
* Life expectancy < 1 year
* Recent myocardial infarction (MI) with ST segment elevation (< 72 hours)
* Left ventricular ejection fraction < 30%
* Clearance della creatinina < 30 ml/min. Further exclusion criteria included bed rest orders, patients in a palliative care setting or with therapy limitations.

Restrictions due to the device were height outside the ranfe of 190cm, weight outside the range of 115kg, pacemakers, other electrical stimulators, or implanted medical pumps.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of LOLE.K reducing ICU and hospital stay | 12 months
  The autors proposal aims to reducing the ICU and Hospital stay in cardiac surgery patients through mobilization and postural drainage. The authors aim to discharge patients from the ICU within two days of surgery and discharge them from the hospital within two weeks.
  Therefore, the unit of measurement is expressed in the number of days elapsed from admission to discharge, both from the intensive care unit and from the hospital overall.
Effectiveness of LOLE.K reducing duration of Mechanical ventilation | 12 months
  One of the primary objectives of this study is to achieve a reduction in the duration of mechanical ventilation compatibly with each patient's specific preoperative and postoperative conditions. In addition to the invasive ventilation phase (ventilator), a reduction in the use of non-invasive ventilation (NIV) is also sought during the immediate postoperative period, up to seven days after surgery.
  The unite of measurement is the number of days the patient requires non-invasive ventilation following extubation.
Effectiveness of LOLE.K enhancing functional outcomes | Maximum 12 months for the entire study, from enrollment to 6 months after discharge
  To assess physical functioning and the associated return to usual activities, the 36-Item Short Form Health Survey version 2 (SF-36 v2) , will be administered 12 weeks after surgery. This questionnaire measures a wide range of symptoms, experiences, and health outcomes across eight domains comprising thirty-six items, addressing gaps in the assessment of patient-reported outcomes throughout the care continuum.
  The unit of measurement is the SF-36 domain score (0-100).
Effectiveness of LOLE.K in patient satisfaction | Maximum 12 months for the entire study, from enrollment to 6 months after discharge
  To characterize patient satisfaction, we will record pain, anxiety, and satisfaction levels during mobilization, all assessed using the Numeric Rating Scale (NRS, 0-10), where 0 indicates no pain and 10 represents the worst pain imaginable. Therefore, the unit of measurement is expressed in points on a 0-10 scale.

SECONDARY OUTCOMES:
Muscular and neurological recovery | Maximum 12 months for the entire study, from enrollment to 6 months after discharge
  Verify the benefits for muscle recovery with the multifunctional bed in patients undergoing cardiac surgery. The authors intend to demonstrate that the bed's special features promote muscle healing process thanks to the programming of cyclical postural transitions specific to cardiac surgery patients. The strength recovery is measured using a dynamometer for Lower limb and Handgrip-Test, evaluating the variation from T0 to T4.
  The unite of measurement for this outcome is Kilogram (Kg).
Neurological and psychological well-being | Maximum 12 months for the entire study, from enrollment to 6 months after discharge
  To assess Neurological and psychological well-being the authors employ 36-Item Short Form Health Survey version 2 (SF-36 v2) 12 weeks after surgery. This questionnaire measures a wide range of symptoms, experiences, and health outcomes across eight domains comprising thirty-six items, addressing gaps in the assessment of patient-reported outcomes throughout the care continuum.
  The unit of measurement is the SF-36 domain score (0-100).
wound healing | 12 months
  One of the objectives of this study is to demonstrate the effectiveness of the LOLE.K bed in wound healing. Through early mobilization of the patient using the cyclical postural changes provided by the multifunctional robotic bed.
  To define the degree of superficial or deep wound infection is used a clinical scoring system (from 0 to 12 points).

CONTACTS AND LOCATIONS:
Locations (1):
- AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno, Campani, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Noss C, Prusinkiewicz C, Nelson G, Patel PA, Augoustides JG, Gregory AJ. Enhanced Recovery for Cardiac Surgery. J Cardiothorac Vasc Anesth. 2018 Dec;32(6):2760-2770. doi: 10.1053/j.jvca.2018.01.045. Epub 2018 Jan 31. PMID 29503121
- [Background] Lay-Ekuakille A, Chiffi C, Celesti A, Rahman MZU, Singh SP. Infrared Monitoring of Oxygenation Process Generated by Robotic Verticalization in Bedridden People. IEEE Sens J. 2021 Mar 25;21(13):14426-14433. doi: 10.1109/JSEN.2021.3068670. eCollection 2021 Jul 1. PMID 35790096